CLINICAL TRIAL: NCT04646434
Title: Investigating the Correlation Between the Brain and Pelvic Floor Muscle Activity of Patients Who Had or Are Undergoing Robot-Assisted Radical Prostatectomy
Brief Title: Brain and Pelvic Floor Muscle Activity of Patients Who Had or Are Undergoing Robot-Assisted Radical Prostatectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: I 822320; NCI-2020-08299 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 822320 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2020-11-04; First posted 2020-11-30 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Neurofeedback; Urodynamics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive Care (brain and muscle monitoring, questionnaire) (Experimental): Patients perform standard of care Kegel exercises while undergoing brain and muscle activity monitoring by UDS, EEG and EMG, respectively, before surgery, 6 weeks after surgery, and at 3, and 6 months after surgery. Patients complete questionnaires over 5-10 minutes about urinary function
  Interventions: Procedure: Electroencephalography; Procedure: Electromyography; Other: Questionnaire Administration; Procedure: Urodynamics (UDS)

INTERVENTIONS:
Procedure: Electroencephalography — Undergo EEG
  Other Names: EEG; electroencephalogram
Procedure: Electromyography — Undergo EMG
  Other Names: EMG
Other: Questionnaire Administration — Complete questionnaire
Procedure: Urodynamics (UDS) — Undergo UDS
  Other Names: UDS

SUMMARY:
This trial investigates brain and pelvic floor muscle activity in patients undergoing robot-assisted radical prostatectomy. This trial may help identify the brain waves that are associated with muscles involved in giving patients control over the bladder.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

* Identify pelvic floor muscle (PFM) activity on electromyogram (EMG) and electroencephalography (EEG).
* Identify any synchrony in EMG and EEG for PFM activity.
* Identify any relationship between EEG activity and UDS findings.

SECONDARY OBJECTIVES:

I. Identify changes in EEG and EMG activity with Kegel exercise. II. Examine relationship between EEG activity and continence.

EXPLORATORY OBJECTIVE:

I. Examine feasibility of replacing EMG with EEG monitoring for muscle activity.

OUTLINE:

Patients perform standard of care Kegel exercises while undergoing brain and muscle activity monitoring by EEG and EMG and UDS, respectively, before surgery, 6 weeks after surgery, 3,months after surgery and 6 months after surgery.. Patients complete questionnaires over 5-10 minutes about urinary function.

ELIGIBILITY:
Inclusion Criteria:

* Adults who had or are undergoing robot-assisted radical prostatectomy (RARP)
* Must be continent preoperatively
* Participant or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Unwilling or unable to follow protocol requirements
* Any condition which in the Investigator's opinion deems the participant an unsuitable candidate for study participation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-07-13 (Actual); Primary Completion 2029-07-13 (Estimated); Study Completion 2029-07-13 (Estimated)

PRIMARY OUTCOMES:
EEG measures obtained during urination. | Up to 6 months after surgery
  Recordings of brain and muscle activity will be collected during urination
Pelvic floor muscle (PFM) EEG measures | Up to 6 months
  Simultaneous recordings of brain activity using electrodes attached to the scalp and muscle activities of muscles of the anal sphincter with electrodes bonded to the skin.
Identification of Areas of synchrony in EEG Patterns and associated Urodynamics (UDS) findings | UP to 6 months
  UDS data of Incontinence/continence will be monitored along with EEG recordings of brain activity during urination.

SECONDARY OUTCOMES:
EEG and EMG biofeedback | Up to 6 months
  Patients will perform Kegel exercises while brain and muscle activity are monitored using a 128-channel EEG headset and up to 24 channel EMG system
Improvement of continence | Throughout life of study up to 6 months after surgery
  International Prostate Symptom score - an 8 question screening tool -with a score from 0= never experienced to 5= almost always experienced.

CONTACTS AND LOCATIONS:
Overall Officials: Khurshid A Guru, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States